CLINICAL TRIAL: NCT05205902
Title: TOtal Skin Electron Beam Therapy (Low-dose) for Tumor Clone Eradication in Early-stage Mycosis Fungoides: a Prospective Randomized Controlled Study
Brief Title: TOtal Skin Electron Beam Therapy (Low-dose) for Tumor Clone Eradication in Early-stage Mycosis Fungoides
Acronym: TOTEM-01
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200128
Record Dates: First submitted 2022-01-24; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Mycosis Fungoides; Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose total-skin electron-beam therapy (Other): Low-dose total skin electron beam therapy (12 Gy) will be delivered to the patient in 4 Gy/week, 1 Gy/day over 3 weeks by symmetrical electron beams of 6 MeV energy via a linac accelerator.
  Interventions: Other: Low-dose total-skin electron-beam therapy
- Phototherapy (Other): Phototherapy will be given 3 times a week during 2 months, then twice a week during one month, then once a week during one month, or until disease progression or unacceptable side effect, whatever comes first.
  Patients with plaques will receive PUVA therapy and patients with patches only will receive narrow-band UVB therapy.
  Interventions: Other: Phototherapy

INTERVENTIONS:
Other: Low-dose total-skin electron-beam therapy — Low-dose total skin electron beam therapy (12 Gy) will be delivered to the patient in 4 Gy/week, 1 Gy/day over 3 weeks by symmetrical electron beams of 6 MeV energy via a linac accelerator.
  Arms: Low-dose total-skin electron-beam therapy
Other: Phototherapy — Phototherapy will be given 3 times a week during 2 months, then twice a week during one month, then once a week during one month, or until disease progression or unacceptable side effect, whatever comes first.
  Patients with plaques will receive PUVA therapy and patients with patches only will receive narrow-band UVB therapy.
  Arms: Phototherapy

SUMMARY:
Primary cutaneous T-cell lymphomas are a group of peripheral T-cell lymphomas that primarily involve the skin. Mycosis fungoides (MF) is the most frequent subtype. Most patients with early-stage MF (i.e., patches and plaques of the skin without extracutaneous involvement) have a good prognosis but a subset of patients progress to incurable advanced-stage disease with an overall survival (OS) less than 5 years and an impaired quality of life.

We have recently identified the tumor clone frequency in lesional skin (measured by high-throughput sequencing of the TCRB locus) as the most important prognostic factor of progression-free survival (PFS) and OS in a retrospective analysis on 210 patients with early-stage MF (p<0.001).

Phototherapy is a standard therapeutic option in early-stage MF but fails to eradicate the tumor clone from the skin.

Low-dose total-skin electron-beam therapy (LDTSEBT, 12 Gy over a 3-week period) has been shown to be safe and highly effective in MF with an 88% overall response rate and a better safety profile compared to standard-dose total-skin electron-beam therapy, in a pooled analysis from 3 phase II trials on 33 patients and a retrospective analysis of 12 patients treated with LDTSEBT.

We hypothesize that the use of LDTSEBT is associated with a significantly higher 1-year PFS compared to conventional treatment with phototherapy. Our secondary hypotheses are that LDTSEBT is associated with a higher tumor T-cell clone eradication compared to phototherapy, and improves OS and quality of life in patients with skin-limited MF.

The main objective of this study is therefore to prospectively determine if LDTSEBT is associated with a higher 1-year progression-free survival in patients with early-stage mycosis fungoides, compared to conventional treatment with phototherapy.

The primary endpoint is PFS at 12 months after study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histopathologically confirmed diagnosis of International Society for Cutaneous Lymphomas (ISCL) / European Organisation for Research and Treatment of Cancer (EORTC) mycosis fungoides stage IB or IIA

Exclusion Criteria:

* Poor performance status: WHO performance status score > 2
* Physically unable to maintain the posture
* Patient with no health coverage
* Patient under guardianship or curatorship
* Previous history of dose-limiting radiation therapy in the field
* Previous history of dose-limiting phototherapy
* Previous history of melanoma, skin squamous cell carcinoma or basal cell carcinoma or other absolute contraindication to phototherapy (including a history of lupus, xeroderma pigmentosum, or porphyria)
* Pregnant or breastfeeding woman
* Contraindication to methoxsalen (severe liver, renal or heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | at 12 months
  Progression will be defined clinically as >25% increase in the modified Severity Weighted Assessment Tool (mSWAT) score from baseline or progression to advanced stage, according to the ISCL/EORTC criteria , or the onset of a new treatment of MF (excepted the use of topical corticosteroids, which is allowed during the study, and will not be considered as a new treatment

SECONDARY OUTCOMES:
Proportion of patients with tumor clone eradication in skin | at 4 months after inclusion
  Tumor clone eradication in skin will be defined by >90% reduction in the tumor cell content (tumor cells/100 ng DNA by high throughput sequencing of TCRB in a lesional skin biopsy) in skin
Complete response rate | at 4 months after inclusion
  Complete response rate will be assessed using ISCL/EORTC criteria
Overall response rates | at 4 months after inclusion
  Overall response rate will be assessed using ISCL/EORTC criteria
Progression-free survival | at 5 years post inclusion
  Progression will be defined clinically as >25% increase in the modified Severity Weighted Assessment Tool (mSWAT) score from baseline or progression to advanced stage, according to the ISCL/EORTC criteria , or the onset of a new treatment of MF (excepted the use of topical corticosteroids, which is allowed during the study, and will not be considered as a new treatment
Overall survival | at 5 years post inclusion
Quality of life as measured by the EORTC QLQ-C30 | at inclusion
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 1 month
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 4 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 1 year
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 2 years
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 3 years
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 4 years
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the EORTC QLQ-C30 | at 5 years
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the Skindex scale | at inclusion
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life as measured by the Skindex scale | at 1 month
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Quality of life as measured by the Skindex scale | at 4 months
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Quality of life as measured by the Skindex scale | at 1 year
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Quality of life as measured by the Skindex scale | at 2 years
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Quality of life as measured by the Skindex scale | at 3 years
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Quality of life as measured by the Skindex scale | at 4 years
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Quality of life as measured by the Skindex scale | at 5 years
  Quality of life will be measured by the Skindex scale-29 instruments which Measure the Effects of Skin Disease on Quality of Life The Skindex-29 scale is a three-dimensional,dermatology-specific health related quality of life (HRQL) questionnaire. thirty items are combined to form three domains: symptoms,emotions, and functioning. The overall score are expressed on a 100-point scale. A higher scores indicate lower level of quality of life.
Proportion of patients with side effects | up to 5 years
  Evaluated by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

IPD SHARING:
Plan to Share IPD: Undecided